CLINICAL TRIAL: NCT02847611
Title: Validation of the Dynamometer LABIN
Acronym: DYNAVAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Department Physical Measures (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0274; 2015-A01732-47 (Other: 2015-A01732-47)
Record Dates: First submitted 2016-07-19; First posted 2016-07-28 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Healthy Volunteers
Keywords: Dynamometer mechanic; Strength of prehension; Comparison; Device; Diagnosis; Healthy Volunteers
MeSH Terms: conditions — Disease

ARMS (2):
- Jamar then Labin (Experimental): The order of the using of the dynamometers "Jamar then Labin" or "Labin then Jamar" is chosen by randomization
  Interventions: Device: Dynamometer LABIN
- Labin then Jamar (Experimental): The order of the using of the dynamometers "Jamar then Labin" or "Labin then Jamar" is chosen by randomization
  Interventions: Device: Dynamometer LABIN

INTERVENTIONS:
Device: Dynamometer LABIN — LABIN is a prototype of dynamometer containing a handle of metal strength, connected with a sensor of pressure registering(recording) the applied strength and transmitting the data in a computer showing an IT curve of the strength according to time.

SUMMARY:
The main objective of this work is to validate the dynamometer LABIN in comparison with the technique of gold-standard reference JAMAR, in a healthy population.

The infringement of the prehension is frequent and impacts on the social and professional quality of life of the patients. There are numerous instruments measuring the strength of prehension. The JAMAR is a mechanical, hydraulic dynamometer, exploring in kilograms the maximal strength of the prehension. It is at present Gold Standard for the measure of the strength of prehension. There is for the moment no electronic known instrument exploring the endurance of the strength of prehension during an effort of tightening. This parameter would indeed be interesting for the exploration in geriatrics and in the neuromuscular pathologies.

This study justifies itself by the fact that the dynamometer LABIN should allow the evaluation of the muscular endurance of the strength of hand as complement of the peak of strength

DETAILED DESCRIPTION:
Measure of the strength of prehension with JAMAR and LABIN according to the following protocol:

* Position: the subject sits comfortably on a chair without armrests, feet put on the ground, the pond at the bottom of the seat, the hips and the knees in 90 ° of flexion, shoulder in adduction and neutral rotation, the elbow bent in 90 °, forearm in neutral position, the wrist between 0 and 30 ° of extension and between 0 and 15 ° of slope ulnaire. The dynamometer is vertically presented and in front of the forearm to maintain the standardized positions.
* Test: regulation of the zero by making a vacuous acquisition during 5 seconds. The order "Jamar then Labin" or Labin then Jamar is chosen by randomization. The operator encourages the subject to every test. The subject does not see the curve displaying.
* Test: 3 clampings of a handle of a dynamometer LABIN by the right hand during 5 seconds, with a break of 30 seconds between the tests. After 2 minutes of break the subjects make 3 clampings with a left hand. After that , the same session is realized with the dynamometer JAMAR

The order "Jamar then Labin" or Labin then Jamar is chosen by randomization. The operator encourages the subject to every test. The subject does not see the curve displaying.

Total duration of participation in the study for the patient: 30 minutes

Main analysis: the calculation of the coefficient of correlation (Pearson or Spearman with regard to the statistical distribution), coefficient of linen concordance and the coefficient of intra-classy correlation.

ELIGIBILITY:
Inclusion Criteria:

* Age : > 20 years and <60 years
* Professionally active
* Right-handed(right-wing) or left-handed person
* Volunteer
* Subjects have given its consent in writing to participate in the study

Exclusion Criteria:

* Subjects with a trauma or surgery of the upper limb
* Subjects with a diabetes
* Subjects with a dysthyroïdie
* Subjects with a neurological disease
* Subjects with a syndrome canalaire of the upper limb
* Subjects with a cutaneous disorders(confusions) of the cognitive upper

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2016-07-08 (Actual); Study Completion 2016-07-08 (Actual)

PRIMARY OUTCOMES:
Measure of the strength of prehension (in Kg). | at day 1
  measure of the strength of prehension in kilogram by using of the JAMAR ( hydraulic dynamometer), and the LABIN (electronic dynamometer provided with a sensor of pressure).

SECONDARY OUTCOMES:
The comfort of the using the dynamometer LABIN | at day 1
  A note of discomfort on Simple Verbal Scale from 0 to 10 (max.) is attributed by the subject
muscular endurance, estimated by dynamometer LABIN preservation of the strength for the LABIN | at day 1
  Change from baselin in measure muscular endurance (The calculation of the horizontal length under the graphic curve which will be exploited by the colleagues of the IUT)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel COUDEYRE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Result] Hamilton GF, McDonald C, Chenier TC. Measurement of grip strength: validity and reliability of the sphygmomanometer and jamar grip dynamometer. J Orthop Sports Phys Ther. 1992;16(5):215-9. doi: 10.2519/jospt.1992.16.5.215. PMID 18796752
- [Result] Harkonen R, Harju R, Alaranta H. Accuracy of the Jamar dynamometer. J Hand Ther. 1993 Oct-Dec;6(4):259-62. doi: 10.1016/s0894-1130(12)80326-7. PMID 8124439
- [Result] Bautmans I, Mets T. A fatigue resistance test for elderly persons based on grip strength: reliability and comparison with healthy young subjects. Aging Clin Exp Res. 2005 Jun;17(3):217-22. doi: 10.1007/BF03324600. PMID 16110735
- [Result] Bellace JV, Healy D, Besser MP, Byron T, Hohman L. Validity of the Dexter Evaluation System's Jamar dynamometer attachment for assessment of hand grip strength in a normal population. J Hand Ther. 2000 Jan-Mar;13(1):46-51. doi: 10.1016/s0894-1130(00)80052-6. PMID 10718222
- [Result] Martin-Ponce E, Hernandez-Betancor I, Gonzalez-Reimers E, Hernandez-Luis R, Martinez-Riera A, Santolaria F. Prognostic value of physical function tests: hand grip strength and six-minute walking test in elderly hospitalized patients. Sci Rep. 2014 Dec 22;4:7530. doi: 10.1038/srep07530. PMID 25531922